CLINICAL TRIAL: NCT03577236
Title: The Zenflow Spring System EU Safety and Performance Study
Acronym: ZEST EU
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zenflow, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLIN-0050
Record Dates: First submitted 2018-05-16; First posted 2018-07-05 (Actual); Last update posted 2021-07-22 (Actual); Status verified 2021-07

CONDITIONS: Benign Prostatic Hyperplasia
MeSH Terms: conditions — Prostatic Hyperplasia

STUDY DESIGN:
Intervention Model Description: Multi-center, prospective, single-arm.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Zenflow Spring System (Experimental): Receives treatment with the investigational device
  Interventions: Device: Zenflow Spring System

INTERVENTIONS:
Device: Zenflow Spring System — The Zenflow Spring System consists of the Spring Delivery System with Implant, Spring Scope, Camera Control Unit (CCU), Measurement Tool, and Spring Retrieval Tool.
  Other Names: Spring Implant

SUMMARY:
The objectives of the trial are to demonstrate the safety and performance of the Zenflow Spring System in relieving the symptoms of obstructive Benign Prostatic Hyperplasia (BPH).

DETAILED DESCRIPTION:
A multi-center, prospective, single arm safety and performance trial. Subjects will be treated either in the Investigator's out-patient treatment room or in the OR, with local anaesthesia only. All subjects will be followed for the entire duration of the study until exit after the 60 month follow-up visit.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is able and willing to comply with all the assessments of the study
2. Patient or patient's legal representative has been informed of the nature of the study, agrees to participate and has signed the informed consent form
3. ≥ 45 years of age
4. Baseline IPSS score > 13, and a baseline Quality of Life (QoL) question score > 3
5. Prostate volume 25 - 80 cc by Trans Rectal Ultrasound (TRUS) or abdominal ultrasound, measured within past 90 days and prostatic urethral length between 2.5- 4.5 cm
6. Failed, intolerant, or patient choice to not take a medication regimen for the treatment of LUTS
7. Patient must meet ONE of the following criteria:

   1. Baseline PSA <= 2.5ng/mL
   2. Baseline PSA >2.5 ng/mL and <=10 ng/mL AND free PSA >=25% of total PSA (no biopsy required or negative biopsy)
   3. Baseline PSA >10ng/mL AND negative prostate biopsy1 result within 12 months
   4. Negative prostate biopsy1 within 12 months if abnormal digital rectal examination
   5. 3 Tesla MRI of the prostate, with normal findings, within 12 months prior to the baseline visit

Exclusion Criteria:

1. Obstructive intravesical median prostatic lobe which, in the opinion of the Investigator, would not benefit from treatment
2. Urethral stricture, meatal stenosis, or bladder neck obstruction - either current, or recurrent requiring 2 or more dilations as reported in the patient's history
3. Requiring self-catheterization to void
4. Baseline PSA > 10 ng/mL or confirmed or suspected prostate cancer
5. Any of the following, taken from a single uroflowmetry reading:

   1. Peak urinary flow rate > 12 ml/second
   2. Post-void residual (PVR) > 250 ml
   3. Peak Urinary flow rate of > 15 ml/second
   4. < 125ml urinary volume voided at baseline (pre-bladder urinary volume of ≥ 150 ml required)
6. Other condition or disease that might cause urinary retention
7. History of other diseases causing voiding dysfunction
8. Concomitant Urinary Tract Infection (UTI) (subject can be enrolled following successful treatment of UTI and a clean urine test), or a history of recurrent or chronic UTIs (defined as 2 or more UTIs in the past 12 months)
9. Concomitant bladder stones
10. Previous pelvic irradiation or radical pelvic surgery
11. Previous prostate surgery, stent implantations, laser prostatectomy, hyperthermia or another invasive treatment to the prostate
12. Chronic prostatitis, or recurring prostatitis within the past 12 months
13. Known allergy to nickel
14. Life expectancy less than 24 months
15. Use of concomitant medications (e.g., anticholinergics, antispasmodics or antidepressants) affecting bladder function
16. Inability to stop taking anticoagulants and/or antiplatelets for at least 3 days prior to the procedure or coumadin for at least 5 days prior to the procedure (low dose aspirin therapy not prohibited)
17. Taking 5-alpha reductase inhibitors within 3 months of pre-treatment (baseline) evaluation unless evidence of same drug dose for at least 6 months with a stable voiding pattern (the drug dose should not be altered or discontinued throughout the study)
18. Taking one of the following within 2 weeks of pre-treatment (baseline) evaluation:

    1. alpha-blockers,
    2. androgens,
    3. anticholinergics, or
    4. cholinergic medication gonadotropin releasing hormonal analogs
19. Taking one of the following within 24 hours of pre-treatment (baseline) evaluation:

    1. phenylephrine, or
    2. pseudoephedrine
20. Future fertility concerns
21. Any severe illness that might prevent study completion or would confound study results

Min Age: 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2019-01-16 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2024-05-30 (Estimated)

PRIMARY OUTCOMES:
Need for urinary catheterization | 7 days after the procedure
  Rate of extended post-operative urinary catheterization
Successful placement of the Zenflow Spring Implant | Day of discharge up to 7 days following device placement
  Successful deployment and procedural success for the Zenflow System to implant the Spring device in the operating room or an out-patient clinical setting.
Effectiveness of the Spring Implant in reducing symptoms of Benign Prostatic Hyperplasia (BPH) using the International Prostate Symptom Score and Quality of Life Score (IPSS+QoL) | Baseline and 3 months
  The patient is asked to respond to 7 questions related to his urinary health using a rating scale of 0 to 5 where zero is excellent and 5 is the worst possible. The responses to the 7 questions are tallied for a total score. In addition the patient is asked 1 question related to his Quality of Life. The possible responses range from 0 to 6 where 0 is the best and 6 is the worst.

SECONDARY OUTCOMES:
Incidence of procedure or device related serious adverse events | Up to 30 days
  Assessment of any device or procedure related Serious Adverse Events (SAE)
Assessment of Sexual Health Assessment: Change in sexual health measured by change in the Sexual Health Inventory for Men (SHIM) questionnaire score | Baseline, 3, 6, 12, & 24 months
  The patient selects the most appropriate response to 5 questions about his sexual health. Each response has an assigned value between 1 and 5. The numeric values are tallied for a total score.
Assessment of Sexual Health Assessment: Change in sexual health measured by change in ability to ejaculate using the Male Sexual Health Questionnaire - Ejaculatory domain (MSHQ-EjD) | Baseline, 3, 6, 12, & 24 months
  The patient selects the most appropriate response to 4 questions about his sexual health specific to ejaculation. Each response has an assigned value between 0 and 5.
Assessment of Pain, evaluated using a Visual Analog Score (VAS) of 1 to 10 | Baseline, 2 weeks, 1 month and 3 months
  Patient describes pain on a Visual Analog Scale (VAS). The scale is a line labeled 1 at the far left indicating minimal pain and 10 on the right, which is maximum pain.
Assessment of Adverse Events | Up to 2 years
  Rate of adverse events related to the procedure or device.
Effectiveness of the Spring Implant in reducing symptoms of Benign Prostatic Hyperplasia (BPH) | Baseline, 2 weeks, 1, 6, 12, 24 months
  The patient is asked to respond to 7 questions related to his urinary health using a rating scale of 0 to 5 where zero is excellent and 5 is the worst possible. The responses to the 7 questions are tallied for a total score. In addition the patient is asked 1 question related to his Quality of Life. The possible responses range from 0 to 6 where 0 is the best and 6 is the worst.
Effectiveness of the Spring Implant in reducing symptoms of Benign Prostatic Hyperplasia (BPH) | Baseline, 2 weeks, 1, 3, 6, 12, 24 months
  Improvement in flow of urine as measured by uroflowmetry machine.
Effectiveness of the Spring Implant in reducing symptoms of Benign Prostatic Hyperplasia (BPH) | Up to 2 years
  Incidence of repeat invasive treatment for Lower Urinary Tract Symptoms (LUTS) or increase in dosage or initiation of new medication to treat symptoms of BPH.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Gilling, MD, Principal Investigator — Tauranga Urology Research Ltd.
Locations (5):
- Australia (4):
  - Australian Clinical Trials, Wahroonga, New South Wales
  - South Coast Urology, Wollongong, New South Wales
  - Goldfields Urology, Bendigo, Victoria
  - Royal Melbourne Hospital, Melbourne, Victoria
- Urology Bay of Plenty, Tauranga, New Zealand

IPD SHARING:
Plan to Share IPD: No